CLINICAL TRIAL: NCT01591746
Title: Botulinum Toxin A in Tissue Expander Breast Reconstruction: A Double-Blinded Randomized Controlled Trial
Brief Title: Botulinum Toxin A (Botox) in Tissue Expander Breast Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Valerie Lemaine, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11-001687
Record Dates: First submitted 2012-04-13; First posted 2012-05-04 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Pain, Postoperative; BRCA1 Mutation; BRCA2 Mutation; Breast Diseases; Neoplasms
Keywords: Mastectomy; Mammaplasty; Breast reconstruction; Tissue expansion; Botulinum toxins, Type A; Quality of Life; Acellular dermal matrix
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Breast Diseases; Neoplasms | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A - Botulinum Toxin Type A (Experimental): 100 Units of Botulinum toxin A diluted in 5 mL 0.9% Sodium Chloride (NaCl) in the pectoralis major muscle in each operated breast
  Interventions: Drug: Botulinum Toxin Type A
- Group B - Placebo (Placebo Comparator): 5 mL 0.9% NaCl injection to the pectoralis major muscle in each operated breast
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Other Names: BOTOX
  Arms: Group A - Botulinum Toxin Type A
Drug: Placebo — 5 mL 0.9% NaCl solution to mimic Botulinum Toxin Type A
  Other Names: Sodium chloride solution
  Arms: Group B - Placebo

SUMMARY:
Each year, the number of breast cancer survivors who choose post-mastectomy breast reconstruction keeps rising. Among women who elect to pursue breast reconstruction, approximately 75% will choose prosthetic breast reconstruction. Implant-based breast reconstruction is frequently achieved in two-stages. The first stage consists of the placement of a tissue expander after mastectomy. This is followed by a period of biweekly tissue expansions that can last several months. In the second stage, the tissue expander is removed in a surgical procedure and replaced with a permanent breast implant. Tissue expansion is a well-established breast reconstruction technique characterized by high success rates and high patient satisfaction. Despite the well-recognized advantages of this successful breast reconstruction technique, the subpectoral placement of a tissue expander is associated with significant pain and discomfort in the immediate post-operative period and during the phase of tissue expansion. Pectoralis major muscle spasm is a frequently reported problem during tissue expansion. Legeby et al. recently showed that women who underwent prosthetic breast reconstruction had higher pain scores and took more analgesics that those who did not choose post-mastectomy reconstruction.

In the past 10 years, publications on the use of botulinum toxin A (BTX-A) for pain relief in a wide array of clinical conditions have increased tremendously. BTX-A is one of the neurotoxins produced by Clostridium botulinum bacteria. By reversibly inhibiting neurotransmitter release, BTX-A has both analgesic and paralytic properties. The analgesic action of BTX-A was initially thought to be related to its effects on muscular contraction. However, a recent in vitro study of embryonic rat dorsal neurons did confirm that BTX-A inhibits release of substance P, a neurotransmitter associated with pain and inflammatory reactions. The presence of analgesic properties of BTX-A is increasingly supported by several clinical observations: pain relief with BTX-A injections has been reported for migraine headaches, chronic pelvic, chronic tennis elbow, and post-operative pain control for lower limb lengthening correction, among others.

This aspect has never been studied in breast cancer survivors who elect to pursue breast reconstruction with tissue expanders. Furthermore, physical function outcomes are important to consider with BTX-A use because the link between temporary muscle paralysis and improvements in participation in daily activities is not a given.

The investigators propose to complete a double-blinded prospective randomized controlled trial of women undergoing unilateral and bilateral mastectomies with immediate placement of tissue expanders, to establish the efficacy and safety of BTX-A in alleviating pain and in improving physical well-being during the expansion period.

DETAILED DESCRIPTION:
Consecutively enrolled eligible women will be randomized into one of two different treatment groups: 1) Group receiving BTX-A, and 2) Group receiving a placebo. All consenting subjects will be randomized to receive either a single injection of 100 units of BTX-A, or a placebo (saline water), during surgery in the pectoralis major muscle on the operated side once the mastectomy and the breast reconstruction have been completed. Expected duration of subject participation is 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years of age, who will undergo immediate unilateral or bilateral tissue expander breast reconstruction following therapeutic skin-sparing or nipple-sparing mastectomy
* Women at least 18 years of age, who will undergo immediate bilateral tissue expanders breast reconstruction following risk-reduction (prophylactic) skin-sparing or nipple-sparing mastectomy

Exclusion Criteria:

* Subjects who are unable to read or speak English
* Breast reconstruction using the latissimus dorsi flap combined with a tissue expander
* Documented diagnosis of chronic pain, upper limb spasticity, cervical dystonia, axillary hyperhidrosis, strabismus or blepharospasm
* Hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation
* Infection at the proposed site of injection
* Pre-existing neuromuscular disorders (including diagnosed myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis)
* Aminoglycosides intake at the time of surgery (these antibiotics can potentiate the effect of BTX-A)
* Women who are pregnant or breast feeding
* Presence of breast implants from previous breast surgery
* Reported use of Botox within 4 months prior to planned surgical date

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Lemaine, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - Botulinum Toxin Type A: 100 Units of Botulinum toxin A diluted in 5 mL 0.9% Sodium Chloride (NaCl) in the pectoralis major muscle in each operated breast
  Botulinum Toxin Type A
Period: Overall Study
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo
Started | 68 | 63
Completed | 68 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo | Total
Number analyzed (Participants) | 68 | 63 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.1) | 48.4 (11.5) | 49.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 63 | 131
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 68 | 63 | 131
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (5.9) | 26.6 (8.1) | 27.1 (7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Pain Scores Using a Numeric Pain Intensity Scale
Description: The numeric pain intensity scale (NPIS) will be completed at the preoperative visit and again at the first postoperative visit. The NPIS is a visual analog scale (VAS) commonly used to assess clinical pain. Subjects are asked to rate their pain on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: preoperative visit, first postoperative visit (1-2 weeks post surgery)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo
Number analyzed (Participants) | 68 | 63
score on a scale | 2 [1.5 to 4] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Group A - Botulinum Toxin Type A vs Group B - Placebo; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Physical Well-Being Using the BREAST-Q, Reconstruction Module
Description: The Physical Well-Being scale of the BREAST-Q, Reconstruction module, will be used for this purpose. The BREAST-Q is a validated patient-reported outcome measure to accurately assess quality of life and patient satisfaction. The Reconstruction module Physical Well-Being scale has questions on the function and participation in activities before and after breast reconstruction. For this study, subjects were asked to answer 16 questions on how often they experienced each symptom, using score of 1 to 5, where 1 was none of the time and 5 was very often. Answers from these questions were combined to provide a total physical well-being score (for a total possible range of 16-80) for each patient at each visit. Lower scores reflected fewer symptoms and higher satisfaction where higher scores reflected more symptoms and less satisfaction.
Time Frame: first post-operative visit (1-2 weeks post surgery)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo
Number analyzed (Participants) | 68 | 63
score on a scale | 63 [57 to 68] | 60 [57 to 68]
Statistical Analysis 1: Comparison: Group A - Botulinum Toxin Type A vs Group B - Placebo; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Initial Intraoperative Fill Volume in Milliliters (mL)
Description: The amount of initial intraoperative fill volume in milliliters (mL) in the tissue expander at the time of surgery divided by the manufacturers recommended total tissue expander volume will be measured. Each breast will be measured separately.
Time Frame: Single intra-operative measurement at first surgery
Population: Volume measurements were not captured for all subjects.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo
Number analyzed (Participants) | 60 | 60
mL
  Right breast | 63.5 (23.0) | 60.4 (20.0)
  Left breast | 60.1 (23.1) | 60.0 (21.1)
Statistical Analysis 1: Comparison: Group A - Botulinum Toxin Type A vs Group B - Placebo; Right breast initial percent volume expansion; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group A - Botulinum Toxin Type A vs Group B - Placebo; Left breast initial percent volume expansion; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Tissue Expansion Visits
Description: The total number of tissue expansion visits completed post-operatively.
Time Frame: up to 24 weeks post-operatively
Measure: Median (Inter-Quartile Range); unit: visits
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo
Number analyzed (Participants) | 66 | 62
visits | 3 [2 to 4] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Group A - Botulinum Toxin Type A vs Group B - Placebo; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Total Volume of Tissue Expansion
Description: Measurement of total expansion volume in milliliters (mL).
Time Frame: Up to 24 weeks post-operatively
Population: Volume measurement were not captured on all subjects.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo
Number analyzed (Participants) | 61 | 59
mL | 80 [63 to 104] | 75 [56 to 100]
Statistical Analysis 1: Comparison: Group A - Botulinum Toxin Type A vs Group B - Placebo; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Rate of Reconstruction Failure
Description: The rate of reconstruction failure will be measured by the number of subjects who have tissue expander removal.
Time Frame: 6 months after first surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo
Number analyzed (Participants) | 68 | 63
Participants | 1 | 0
Statistical Analysis 1: Comparison: Group A - Botulinum Toxin Type A vs Group B - Placebo; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until four months postoperatively for each subject, a total average of five years.
Arm/Group | Group A - Botulinum Toxin Type A | Group B - Placebo
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/63
Other Adverse Events (participants affected / at risk) | 15/68 | 14/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Botulinum Toxin Type A (N=68) | Group B - Placebo (N=63)
Surgical site infection (Infections and infestations) | 1 (1) | 2 (2)
Hematoma requiring reoperation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Seroma (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Mastectomy skin flap necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Delayed wound healing (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Unplanned reoperation (Surgical and medical procedures) | 7 (7) | 4 (4)

LIMITATIONS AND CAVEATS:
A practice change from patients receiving paravertebral blocks preoperatively to intraoperative field blocks with liposomal bupivacaine;data not collected on postoperative oral narcotic consumption;study designed to detect 25% decrease in pain score.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT01591746/Prot_SAP_000.pdf